# Healthcare resource utilisation, common mental health problems, and infections in people with inflammatory bowel disease (IBD)

**NCT number:** Not available at submission

**Document date:** 6th Dec 2018

# **Academic contributors**

Dr Kevin Barrett<sup>1</sup>, Dr Peter Irving<sup>2</sup>, Professor Simon de Lusignan<sup>3, 4</sup>

- <sup>1</sup> New Road Surgery, Croxley Green, Hertfordshire, UK
- <sup>2</sup> Department of Gastroenterology, Guy's & St Thomas' Hospital, London, UK.
- <sup>3</sup> Department of Clinical and Experimental Medicine, University of Surrey, Guildford, United Kingdom
- <sup>4</sup> Royal College of General Practitioners, London, UK

The research is supported by Momentum Data Ltd



# **Abstract**

#### **Background**

Ulcerative colitis (UC) and Crohn's disease (CD) are chronic inflammatory conditions collectively termed inflammatory bowel disease (IBD). Both conditions are chronic and involve a lifetime of treatment. Current treatment strategies for IBD focus on the use of immune modulating medications, which have the potential to increase the risk of common infections. An understanding of the healthcare resource utilisation and overall infection risk in IBD is therefore important. Despite increasing treatment options, quality of life is significantly reduced in people with IBD and a high prevalence of mental health disorders has been reported. However, the magnitude of any potential association between IBD and mental illness in adults has not yet been fully explored.

#### **Objective**

We aim to provide an accurate and contemporary measurement of the current healthcare resource utilisation in people with IBD. We also aim to provide estimates of infection incidence in this population and the prevalence of common mental health conditions. We will also

#### Method

We will identify UC and CD using algorithms validated for accurately identifying these conditions from primary care records in the UK. We will identify a prevalent cohort of adults with IBD with the RCGP RSC network over the last decade. We will identify a matched cohort of people without IBD; matched on age, gender and primary care practice. Across these cohorts we will compare healthcare resource utilisation (primary care attendances, number of primary care prescriptions for antidepressant and anxiolytic medications, number of primary care prescriptions for medications used in IBD, recorded secondary care attendances, and issue of statements of fitness for work), incident infections (any common infection, any viral infection, or any gastrointestinal infection), and common mental health conditions (depression, anxiety, and attention deficit hyperactivity disorder).

# **Lay Summary**

Ulcerative colitis and Crohn's disease are the commonest types of inflammatory bowel disease (IBD). Both conditions range in severity from no symptoms to being potentially fatal. Both conditions are treated with medications which supress the immune system. It is not known whether this increases the risk for infections in these conditions. It is also recognised by healthcare professionals that these conditions cause a considerable amount of psychological distress. However, this has never been measured in a large population sample.

These studies will investigate any associations with treatment and new onset infections. They will also examine the relationship between IBD and common mental health problems (specifically, depression and anxiety) and the impact that these have on the healthcare use (including number of GP appointments, hospital attendances, and medication prescriptions. Combined, these studies should provide a better understanding of the impact of IBD on affected people and provide evidence to support the correct allocation of healthcare resources.

# Introduction

Ulcerative colitis (UC) and Crohn's disease (CD) are chronic inflammatory conditions collectively termed inflammatory bowel disease (IBD).¹ In both conditions there is a spectrum of disease ranging from a quiescent state with few or no symptoms to potentially fatal disease. Both conditions commonly require extensive medical intervention over many decades of disease and may also require substantial surgical treatment.², ³ With the global burden of IBD rising, calls have been made for improved treatment options,⁴ and these been met with the development of a range of biologic therapies.¹

Current treatment strategies for UC focus on the use of immune modulating medications. Whilst frequently effective for disease control, these treatments have the potential to increase the risk of common infections,<sup>5, 6</sup> which includes both common and atypical pathogens.<sup>6</sup> An understanding of the infection risk in a community-based population with UC is therefore important. However, the existing literature on infection rates in people with UC has focused almost exclusively on secondary care populations. It therefore remains unclear what the total burden of infectious disease is in a population-based cohort with UC and how this compares to those without UC.

Despite increasing treatment options, quality of life is significantly reduced in people with IBD<sup>7</sup> and the prevalence of mental health disorders has been reported to be higher in children with IBD.<sup>8</sup> However the magnitude of any potential association between IBD and mental illness in adults has not yet been fully explored.

Given the prolonged course of medical treatment in IBD, it is important for payers to have a good understanding of the total healthcare utilisation of people with IBD. Again, in this area, existing studies have focussed on secondary care based cohorts. Little is known about healthcare resource utilisation in primary care, in people with IBD, in the UK.

#### **Aims**

- We aim to describe the incidence of common infections in a population of individuals with IBD, compared to a matched control population without IBD. We will explore all common infections and also focus on viral and gastrointestinal infections.
- 2. We will explore how incidence of infection varies by age, and other factors associated with risk of infection in IBD including medication use.
- 3. We aim to describe the prevalence of common mental health conditions (anxiety, depressive episodes, and recurrent depressive disorder) in people with IBD when compared to an age and gender matched cohort.
- 4. We aim to explore healthcare utilisation in individuals with IBD with and without common mental health problems.

# **Methods**

## Study design

We aim to perform a retrospective matched cohort study. We will match people with UC and CD, to people without IBD. A history of common mental health conditions was assessed at baseline (matching date) in both cohorts, and compared. Both cohorts will be followed-up (retrospectively) from the matching date for incident infections, and healthcare resource utilisation.

#### Data source

We aim to use the Royal College of General Practitioners (RCGP) Research and Surveillance Centre (RSC) database. This database contains the pseudonymised primary care records of the registered population all from a network of GP practices which provide a representative sample of the UK population. The RCGP RSC database contains complete data on all events and clinical entities coded in UK primary care. These include demographic information, clinical diagnoses, laboratory test results, primary care issued prescriptions, process of care codes (e,g. specialist referrals), and anthropometric measurements (e.g., body mass index; BMI), and are coded using the Read coding system. The second system of the provided system of the provided system.

UK general practice records provide several advantages for this study type;<sup>11, 12</sup> UK primary care is a registration-based system (a patient can only register with a single GP), records have been computerised since the 1990s, and pay-for-performance targets (introduced in 2004 through The Quality and Outcomes Framework; QOF) have resulted in consistent high-quality clinical data entry about chronic disease. Studies using the RCGP RSC data have been published across a range of chronic diseases. <sup>13-15</sup> RCGP RSC practices get feedback on their data quality, including using a dashboard. A particular emphasis of this feedback is "episode typing" – designating cases first, new, or ongoing – which helps differentiate incidence from prevalence. <sup>16</sup>

# Study population and outcome measures

All adults (aged ≥18) registered with a GP practice contributing to the RCGP RCS at the time of data extraction will be eligible for inclusion.

#### Definition of the IBD cohort

All individuals with one or more diagnostic codes for UC or CD prior to the study start date were eligible for inclusion in the IBD cohort. The use of diagnostic codes to identify IBD from UK primary care records has been validated and shown to be accurate and to correctly differentiate between UC and CD.<sup>17, 18</sup> The Read codes used to identify UC and CD were based on the codes list used by Abrahami et al.,<sup>18</sup> and mapped to both Read code versions used within the RCGP RSC network (Appendix 1). The use of diagnostic codes to identify IBD has also been shown to have good validity in US claims databases.<sup>19</sup>

#### Definition of the matched cohort

The matched unexposed cohort will be identified by matching individuals with IBD to people without IBD. Matching will be performed on age and gender as a minimum. Follow-up for each matched individual will begin at the same baseline date as those with IBD.

#### Infections outcomes

Infections outcomes will comprise:

- 1. The time to first recorded presentation with a new episode of any common infection during the study period; a composite of upper respiratory tract infections, pneumonia, bronchitis, influenza-like illness, skin infections, genital infections, urinary tract infections and gastrointestinal infections.
- 2. The time to first recorded presentation with a new episode of any viral infection.
- 3. The time to first recorded presentation with a new episode of any episode of gastrointestinal infection.

The Read codes used to identify infections will be adapted from the validated indicators used in routine surveillance by the RCGP RSC. The chosen infections in the composite infections outcomes were selected principally as they represent the majority of the primary care adult infectious disease burden, and include a mixture of viral, bacterial and fungal infections. First or new episodes of an infection are coded accordingly in the database, enabling differentiation from chronic infections or follow-up visits for the same episode. If available, we will also explore type and pathogens contributing to the incident infections.

## Mental health outcomes

The presence of common mental health conditions at baseline will be determined for the case and control cohorts. We will examine three groups of common mental illness as defined by the International Statistical Classification of Diseases and Related Health Problems 10th Revision (ICD10) classification;<sup>20</sup> depressive episodes (F32), recurrent depressive disorder (F33), and non-phobia related anxiety disorders (F41). These conditions are chosen as they represent the most common mental health conditions presenting to primary care.<sup>21</sup> These conditions will be identified using algorithms validated in UK primary care.<sup>22</sup> We selected the algorithms used here (Appendix 2) to optimise the positive predictive value. In brief, we will use a concurrent diagnosis and treatment code to identify acute episodes (depressive episodes and anxiety episodes) and for recurrent depression either a historical code for any depression and current treatment or a recurrent

depression specific diagnosis code (Appendix 2). As a secondary analysis we will also explore the prevalence of attention deficit hyperactivity disorder (ADHD) in the case and control cohorts.

#### Healthcare utilisation outcomes

The components of healthcare utilisation to be examined comprise; number and duration of primary care attendances, number of primary care prescriptions for antidepressant and anxiolytic medications, number of primary care prescriptions for medications used in IBD, recorded secondary care attendances, and issue of statements of fitness for work (also termed fit notes or sick notes).

Antidepressant medication classes to be examined comprise, selective serotonin reuptake inhibitors (SSRIs) and related medications (serotonin and norepinephrine reuptake inhibitors; SNRIs), tricyclic antidepressants (TCAs) and related medications (tetracyclic antidepressant TeCAs), and monoamine oxidase inhibitors (MOAIs). Anxiolytic medications to be examined comprise all benzodiazepines and other related medications indicated for use in anxiety states (Appendix 3). Medications used for the treatment of IBD to be examined will comprise; topical 5-aminosalicylic acid (5-ASA) medications, topical glucocorticoids, oral 5-ASA medications, oral glucocorticoids, non-biologic immunosuppressant medications (cyclosporine, azathioprine, mercaptopurine, methotrexate), and biologic therapies (Appendix 3).

#### Other baseline measures

Socioeconomic status will be defined using the official national measure; the index of multiple deprivation (IMD).<sup>23</sup> This is calculated at the point of data extraction, using patient postcode, with the resultant scores stratified by deprivation quintile. Ethnicity will be extracted from the primary care record and grouped into major ethnic groups; white, black, Asian, mixed, and others.<sup>24</sup> BMI will be defined as the most recently recorded measurement prior to the study start date. Smoking status will be defined using the most recently recorded data prior to the study start date. Diagnosis codes will be used to define the presence of comorbidities at baseline; diabetes, hypertension, atrial fibrillation, angina, myocardial infarction, congestive heart failure, stroke, transient ischaemic attack, chronic kidney disease (stages 3–5), dementia, rheumatoid arthritis, chronic liver disease, asthma and chronic obstructive pulmonary disease (COPD).

# **Statistical Analyses**

#### Comparison of the prevalence of mental health conditions

We will compare the prevalence of the three common mental health conditions in people with IBD and matched controls prior to the baseline date (January 1, 2015). We will stratify groups by age, and gender, and for those with IBD by condition (UC or CD) and duration of disease, and other important baseline factors. We will evaluate differences in baseline characteristics between the cohorts using the  $\chi^2$  test for categorical variables and the unpaired t-test for continuous data. Other statistical tests may be used if appropriate, depending on the data type and distribution.

### Comparison of healthcare utilisation

We will compare the measures of healthcare utilisation between people with IBD and matched cohorts over a follow-up period. Follow-up will end at the earliest of; the study end-date (data extraction date), the date of patient transfer from an included practice, or date of death. All individuals contributing at least 1 day of follow-up will be included for analysis. We will stratify and compare healthcare utilisation in people with IBD by age and gender, condition (UC or CD), duration of disease, the presence of mental health conditions, and other important

confounders. All utilisation outcomes will be adjusted for the duration of followup and reported as event rates.

Where sample size allows we will examine factors associated with increased healthcare utilisation. We will use regression analyses to assess potential associations between healthcare utilisation outcome measures and important patient and treatment factors.

#### Comparison of infections

Infection incidence rates will be calculated as the number of events divided by the total person-years of follow-up and expressed as the number per 1000 person-years. We will estimate the risk of infection in people with and without IBD using Cox proportional hazards models, and report estimated hazard ratios for associations with 95% confidence intervals. We will evaluate factors associated with an increased risk of infection. Factors assessed will include age, gender, socioeconomic status, household size (if available), comorbidities, and UC medications.

All statistical analyses will be performed in the R statistical package.

# **Ethical approval**

Study approval will be requested from the Research Committee of the RCGP RSC. The study does not meet the requirements for formal ethics board review as defined using the NHS Health Research Authority research decision tool (http://www.hra-decisiontools.org.uk/research/).

# **Contributors**

Research support for this project in several areas including data analysis, literature searching, and medication writing will be provided by Momentum Data. John Dennis and Andrew McGovern of Momentum Data have contributed to the writing of this protocol and to the study design. Funding for these studies has been provided by Pfizer UK.

# Scientific rigor and study registration

The team ethos at Momentum Data is to support the highest quality research, for patient benefit, with rigorous scientific standards. Publication bias remains an issue in observational studies. Therefore, if approval is granted the protocol will be registered as an observational study with ClinicalTrials.gov and made publicly available prior to the commencement of data analysis. Any protocol amendments will be published alongside this public record of the study and will be noted in any final publication with the rationale for the modification. Any changes will be assessed for the need for ethics approval and further RCGP RSC study approval; these will be sought if required.

## References

- 1. Baumgart DC, Sandborn WJ. Inflammatory bowel disease: clinical aspects and established and evolving therapies. *The Lancet* 2007; **369**(9573): 1641-57.
- 2. Bodger K. Cost of illness of Crohn's disease. *PharmacoEconomics* 2002; **20**(10): 639-52.
- 3. Bassi A, Dodd S, Williamson P, Bodger K. Cost of illness of inflammatory bowel disease in the UK: a single centre retrospective study. *Gut* 2004; **53**(10): 1471-8.
- 4. Ng SC, Shi HY, Hamidi N, et al. Worldwide incidence and prevalence of inflammatory bowel disease in the 21st century: a systematic review of population-based studies. *The Lancet* 2017; **390**(10114): 2769-78.
- 5. Kucharzik T, Maaser C. Infections and Chronic Inflammatory Bowel Disease. *Viszeralmedizin* 2014; **30**(5): 326-32.
- 6. Toruner M, Loftus EV, Jr., Harmsen WS, et al. Risk factors for opportunistic infections in patients with inflammatory bowel disease. *Gastroenterology* 2008; **134**(4): 929-36.
- 7. Romberg-Camps MJL, Bol Y, Dagnelie PC, et al. Fatigue and health-related quality of life in inflammatory bowel diseaseResults from a population-based study in the Netherlands: The IBD-South Limburg cohort. *Inflammatory Bowel Diseases* 2010; **16**(12): 2137-47.
- 8. Engström I. Mental Health and Psychological Functioning in Children and Adolescents with Inflammatory Bowel Disease: a Comparison with Children having Other Chronic Illnesses and with Healthy Children. *Journal of Child Psychology and Psychiatry* 1992; **33**(3): 563-82.
- 9. Correa A, Hinton W, McGovern A, et al. Royal College of General Practitioners Research and Surveillance Centre (RCGP RSC) sentinel network: a cohort profile. *BMJ open* 2016; **6**(4): e011092.
- 10. de Lusignan S, Liaw ST, Michalakidis G, Jones S. Defining datasets and creating data dictionaries for quality improvement and research in chronic disease using routinely collected data: an ontology-driven approach. *Informatics in primary care* 2011; **19**(3): 127-34.

- 11. de Lusignan S, van Weel C. The use of routinely collected computer data for research in primary care: opportunities and challenges. *Family practice* 2006; **23**(2): 253-63.
- 12. de Lusignan S, Metsemakers JF, Houwink P, Gunnarsdottir V, van der Lei J. Routinely collected general practice data: goldmines for research? A report of the European Federation for Medical Informatics Primary Care Informatics Working Group (EFMI PCIWG) from MIE2006, Maastricht, The Netherlands. *Informatics in primary care* 2006; **14**(3): 203-9.
- 13. Williams R, Alexander G, Armstrong I, et al. Disease burden and costs from excess alcohol consumption, obesity, and viral hepatitis: fourth report of the Lancet Standing Commission on Liver Disease in the UK. *Lancet (London, England)* 2018; **391**(10125): 1097-107.
- 14. Kumar S, de Lusignan S, McGovern A, et al. Ischaemic stroke, haemorrhage, and mortality in older patients with chronic kidney disease newly started on anticoagulation for atrial fibrillation: a population based study from UK primary care. *BMJ (Clinical research ed)* 2018; **360**: k342.
- 15. Woodmansey C, McGovern AP, McCullough KA, et al. Incidence, Demographics, and Clinical Characteristics of Diabetes of the Exocrine Pancreas (Type 3c): A Retrospective Cohort Study. *Diabetes care* 2017; **40**(11): 1486-93.
- 16. Pathirannehelage S, Kumarapeli P, Byford R, Yonova I, Ferreira F, de Lusignan S. Uptake of a Dashboard Designed to Give Realtime Feedback to a Sentinel Network About Key Data Required for Influenza Vaccine Effectiveness Studies. *Stud Health Technol Inform* 2018; **247**: 161-5.
- 17. Stapley SA, Rubin GP, Alsina D, Shephard EA, Rutter MD, Hamilton WT. Clinical features of bowel disease in patients aged <50 years in primary care: a large case-control study. *The British journal of general practice: the journal of the Royal College of General Practitioners* 2017; **67**(658): e336-e44.
- 18. Abrahami D, Douros A, Yin H, et al. Dipeptidyl peptidase-4 inhibitors and incidence of inflammatory bowel disease among patients with type 2 diabetes: population based cohort study. *BMJ* 2018; **360**.
- 19. Ananthakrishnan AN, Cai T, Savova G, et al. Improving case definition of Crohn's disease and ulcerative colitis in electronic medical records using natural language processing: a novel informatics approach. *Inflamm Bowel Dis* 2013; **19**(7): 1411-20.
- 20. World Health Organisation. International Statistical Classification of Diseases and Related Health Problems 10th Revision2016. <a href="http://apps.who.int/classifications/icd10/browse/2016/en">http://apps.who.int/classifications/icd10/browse/2016/en</a> (accessed.
- 21. Kessler RC, Chiu WT, Demler O, Merikangas KR, Walters EE. Prevalence, severity, and comorbidity of 12-month DSM-IV disorders in the National Comorbidity Survey Replication. *Archives of general psychiatry* 2005; **62**(6): 617-27.
- 22. John A, McGregor J, Fone D, et al. Case-finding for common mental disorders of anxiety and depression in primary care: an external validation of routinely collected data. *BMC Medical Informatics and Decision Making* 2016; **16**(1): 35.
- 23. Department for Communities and Local Government. The English Indices of Deprivation. 2015.2015. https://www.gov.uk/government/statistics/english-indices-of-deprivation-2015 (accessed.

24. Tippu Z, Correa A, Liyanage H, et al. Ethnicity Recording in Primary Care Computerised Medical Record Systems: An Ontological Approach. *Journal of innovation in health informatics* 2017; **23**(4): 920.

# **Appendices**

# Appendix 1

| Ulcerative colitis | | |
|---|---|---|
| Read V2 Code | Term<br>ID | Description |
| J41 | All | Ulcerative colitis and/or proctitis |
| J410. | All | Ulcerative proctocolitis |
| J4100 | All | Ulcerative ileocolitis |
| J4101 | All | Ulcerative colitis |
| J4102 | All | Ulcerative rectosigmoiditis |
| J4103 | All | Ulcerative proctitis |
| J4104 | All | Exacerbation of ulcerative colitis |
| J410z | All | Ulcerative proctocolitis NOS |
| J411. | All | Ulcerative (chronic) enterocolitis |
| J412. | All | Ulcerative (chronic) ileocolitis |
| J413. | All | Ulcerative pancolitis |
| N0454 | All | Juvenile arthritis in ulcerative colitis |
| N0310 | All | Arthropathy in ulcerative colitis |
| Read CTV3 | Term | |
| Code | ID | Description |
| XE0ag | All | Ulcerative colitis |
| XaZ2j | All | Left sided ulcerative colitis |
| XaYzX | All | Ulcerative pancolitis |
| XaK6E | All | Exacerbation of ulcerative colitis |
| J410. | All | Ulcerative proctocolitis |
| J4100 | All | Ulcerative ileocolitis |
| J410z | All | Ulcerative proctocolitis NOS |
| Jyu41 | All | [X]Other ulcerative colitis |
| Crohn's disease | <u> </u> | |
| Read V2 Code | Term<br>ID | Description |
| J40 | All | Regional enteritis- Crohn's disease |
| J400. | All | Regional enteritis of the small bowel |
| J4002 | All | Crohn's disease of the termnal ileum |
| J4003 | All | Crohn's disease of the ileum unspecified |
| J4004 | All | Crohn's disease of the ileum NOS |
| J4005 | All | Exacerbation of Crohn's disease of small intestine |
| J400z | All | Crohn's disease of the small bowel NOS |
| J40 | All | Crohn's disease |
| J4012 | All | Exacerbation of Crohn's disease of large intestine |
| J401z | All | Crohn's disease of the largel bowel NOS |
| J402. | All | Regional ileocolitis |
| J40z. | All | Crohn's disease NOS |

| Read CTV3<br>Code | Term<br>ID | Description |
|---|---|---|
| XE2QL | All | Crohn's disease |
| Xa0lh | All | Regional enteritis |
| X302r | All | Crohn's jejunitis |
| X302t | All | Crohn's ileitis |
| J4003 | All | Crohn's disease of the ileum unspecified |
| J4004 | All | Crohn's disease of the ileum NOS |
| J4002 | All | Crohn's disease of terminal ileum |
| J400. | All | Regional enteritis of small bowel |
| XaK6C | All | Exacerbation of Crohn's disease of small intestine |
| J400z | All | Crohn's disease of the small bowel NOS |
| J401. | All | Regional enteritis of the large bowel |
| XE0af | All | Crohn's disease of the large bowel NOS |
| XaK6D | All | Exacerbation of Crohn's disease of large intestine |
| J40z. | All | Regional enteritis NOS |
| J4010 | All | Crohn's colitis |
| J4011 | All | Crohn's proctitis |
| X3050 | All | Perianal Crohn's disease |
| Jyu40 | All | [X]Other Crohn's disease |

**Supplementary table S1.** Read codes used to identify inflammatory bowel disease

# Appendix 2

| Clinical entity | ICD 10 code | Definition |
|---|---|---|
| Anxiety | F41 | Any coded anxiety episode AND concurrent |
| | | treatment for anxiety |
| Depressive episode | F32 | Any coded depressive episode AND |
| | | concurrent treatment for depression |
| Recurrent | F33 | (Any historical code* for a depressive |
| depressive disorder | | episode AND current treatment for |
| | | depression) OR Any code for recurrent |
| | | depressive disorder |
| Anxiety treatments | NA | SSRIs, anxiolytics, counselling, CBT, and |
| | | psychotherapy |
| Depression | NA | SSRIs, TCAs, MAOIs, counselling, CBT, and |
| treatments | | psychotherapy |

**Supplementary table S2.** Algorithms used to identify anxiety episodes, depression episodes, and recurrent major depression. Expressions in capitals equate to Boolean expressions. \*More than 1 year ago. SSRIs = selective serotonin reuptake inhibitors, TCA = tricyclic antidepressants, MAOI = monoamine oxidase inhibitors, CBT = cognitive behavioural therapy.

| Read V2 Code | Term ID | Description |
|--------------|---------|-------------------------------------------------|
| E200. | All | Anxiety states |
| E2000 | All | Anxiety state unspecified |
| E2001 | All | Panic disorder |
| E2002 | All | Generalised anxiety disorder |
| E2003 | All | Anxiety with depression |
| E2004 | All | Chronic anxiety |
| E2005 | All | Recurrent anxiety |
| E200z | All | Anxiety state NOS |
| Eu41. | All | [X]Other anxiety disorders |
| Eu410 | All | [X]Panic disorder [episodic paroxysmal anxiety] |
| Eu411 | All | [X]Generalized anxiety disorder |
| Eu412 | All | [X]Mixed anxiety and depressive disorder |
| Eu413 | All | [X]Other mixed anxiety disorders |
| Eu41y | All | [X]Other specified anxiety disorders |
| Eu41z | All | [X]Anxiety disorder, unspecified |
| Read CTV3 | | |
| Code | Term ID | Description |
| E200. | All | Anxiety disorder |
| XE1Y7 | All | Panic disorder |
| Eu410 | All | [X]Panic disorder [episodic paroxysmal anxiety] |
| E2002 | All | Generalised anxiety disorder |
| X00Sb | All | Mixed anxiety and depressive disorder |
| X00RP | All | Organic anxiety disorder |
| E2004 | All | Chronic anxiety |
| E2005 | All | Recurrent anxiety |
| E200z | All | Anxiety state NOS |
| X00Sc | All | Anxiety hysteria |
| Eu41. | All | [X]Other anxiety disorders |
| Eu413 | All | [X]Other mixed anxiety disorders |
| Eu41z | All | [X]Anxiety disorder, unspecified |

**Supplementary table S3.** Read codes used to identify anxiety episodes.

| Read V2 | Term | |
|---|---|---|
| Code | ID | Description |
| E0013 | All | Presenile dementia with depression |
| E0021 | All | Senile dementia with depression |
| E112. | All | Single major depressive episode |
| E1120 | All | Single major depressive episode, unspecified |
| E1121 | All | Single major depressive episode, mild |
| E1122 | All | Single major depressive episode, moderate |
| | | Single major depressive episode, severe, without mention of |
| E1123 | All | psychosis |
| E1124 | All | Single major depressive episode, severe, with psychosis |
| E1125 | All | Single major depressive episode, in partial or unspecified remission |
| E1126 | All | Single major depressive episode, in full remission |
| E112z | All | Single major depressive episode NOS |
| E113. | All | Recurrent major depressive episode |
| E1130 | All | Recurrent major depressive episodes, unspecified |
| E1131 | All | Recurrent major depressive episodes, mild |
| E1132 | All | Recurrent major depressive episodes, moderate |
| | | Recurrent major depressive episodes, severe, without mention of |
| E1133 | All | psychosis |
| E1134 | All | Recurrent major depressive episodes, severe, with psychosis |
| E1137 | All | Recurrent depression |
| E113z | All | Recurrent major depressive episode NOS |
| E118. | All | Seasonal affective disorder |
| E11y2 | All | Atypical depressive disorder |
| E11z2 | All | Masked depression |
| E130. | All | Reactive depressive psychosis |
| E135. | All | Agitated depression |
| E2003 | All | Anxiety with depression |
| E291. | All | Prolonged depressive reaction |
| E2B | All | Depressive disorder NEC |
| E2B1. | All | Chronic depression |
| E2B0. | All | Postviral depression |
| Eu204 | All | [X]Post-schizophrenic depression |
| Eu251 | All | [X]Schizoaffective disorder, depressive type |
| Eu32. | All | [X]Depressive episode |
| Eu320 | All | [X]Mild depressive episode |
| Eu321 | All | [X]Moderate depressive episode |
| Eu322 | All | [X]Severe depressive episode without psychotic symptoms |
| Eu323 | All | [X]Severe depressive episode with psychotic symptoms |
| Eu324 | All | [X]Mild depression |
| Eu325 | All | [X]Major depression, mild |
| Eu326 | All | [X]Major depression, moderately severe |
| Eu327 | All | [X]Major depression, moderately severe [X]Major depression, severe without psychotic symptoms |
| Eu328 | All | [X]Major depression, severe with psychotic symptoms |

| Eu32y | All | [X]Other depressive episodes |
|---|---|---|
| Eu32z | All | <del> • •</del> |
| | | [X]Depressive episode, unspecified |
| Eu33. | All | [X]Recurrent depressive disorder |
| Eu330 | All | [X]Recurrent depressive disorder, current episode mild |
| Eu331 | All | [X]Recurrent depressive disorder, current episode moderate |
| Eu332 | All | [X]Recurrent depressive disorder, current episode severe without psychotic symptoms |
| EU332 | All | [X]Recurrent depressive disorder, current episode severe with |
| Eu333 | All | psychotic symptoms |
| Eu334 | All | [X]Recurrent depressive disorder, currently in remission |
| Eu33y | All | [X]Other recurrent depressive disorders |
| Eu33z | All | [X]Recurrent depressive disorder, unspecified |
| Eu332<br>Eu412 | All | [X]Mixed anxiety and depressive disorder |
| Read CTV3 | Term | [A] Mixed anxiety and depressive disorder |
| Code | ID | Description |
| X00Sb | All | Mixed anxiety and depressive disorder |
| X00SO | All | Depressive disorder |
| X761L | All | Seasonal affective disorder |
| Xa0wV | All | Recurrent brief depressive disorder |
| X00SQ | All | Agitated depression |
| XE1YC | All | Reactive depression |
| X00SR | All | Endogenous depression |
| X00SS | All | Endogenous depression first episode |
| XE1Y0 | All | Single major depressive episode |
| E1120 | All | Single major depressive episode, unspecified |
| E1120 | All | Single major depressive episode, unspecified |
| E1120 | All | Single major depressive episode, mild |
| E1121<br>E1122 | All | |
| E1122 | All | Single major depressive episode, moderate Single major depressive episode, severe, without mention of |
| E1123 | All | psychosis |
| E1124 | All | Single major depressive episode, severe, with psychosis |
| | 1 1 1 1 1 | Single major depressive episode, severe, with psychosis, psychosis |
| XaX53 | All | in remission |
| E1125 | All | Single major depressive episode, in partial or unspecified remission |
| E1126 | All | Single major depressive episode, in full remission |
| E112z | All | Single major depressive episode NOS |
| XM1GC | All | Endogenous depression - recurrent |
| E1130 | All | Recurrent major depressive episodes, unspecified |
| E1131 | All | Recurrent major depressive episodes, mild |
| E1132 | All | Recurrent major depressive episodes, moderate |
| | | Recurrent major depressive episodes, severe, without mention of |
| E1133 | All | psychosis |
| E1134 | All | Recurrent major depressive episodes, severe, with psychosis |
| 74467 | 433 | Recurrent major depressive episodes, in partial or unspecified |
| E1135 | All | remission |
| E1136 | All | Recurrent major depressive episodes, in full remission |
| E113z | All | Recurrent major depressive episode NOS |

| X00SU | All | Masked depression |
|---|---|---|
| E11y2 | All | Atypical depressive disorder |
| X00S8 | All | Post-schizophrenic depression |
| XSEGJ | All | Major depressive disorder |
| XSKr7 | All | Cotard syndrome |
| XSGol | All | Moderate major depression |
| XSGok | All | Mild major depression |
| XSGom | All | Severe major depression without psychotic features |
| XSGon | All | Severe major depression with psychotic features |
| E1137 | All | Recurrent depression |
| E130. | All | Reactive depressive psychosis |
| E2B | All | Depressive disorder NEC |
| E2B0. | All | Postviral depression |
| E2B1. | All | Chronic depression |
| Eu320 | All | [X]Mild depressive episode |
| Eu321 | All | [X]Moderate depressive episode |
| Eu331 | All | [X]Recurrent depressive disorder, current episode moderate |
| XE1Y1 | All | Recurrent major depressive episodes |
| XE1ZY | All | [X]Severe depressive episode without psychotic symptoms |
| XE1ZZ | All | [X]Severe depressive episode with psychotic symptoms |
| XE1Za | All | [X]Other depressive episodes |
| XE1Zb | All | [X]Depressive episode, unspecified |
| XE1Zd | All | [X]Recurrent depressive disorder, current episode severe without psychotic symptoms |
| XE1Ze | All | [X]Recurrent depressive disorder, current episode severe with |
| XE1Ze<br>XE1Zf | All | psychotic symptoms [VID assument depressive disorder unappedicted] |
| | | [X]Recurrent depressive disorder, unspecified |
| XaB9J | All | Depression NOS |
| XaCHr | All | [X] Single episode agitated depression without psychotic symptoms |
| XaCHs | All | [X] Single episode major depression without psychotic symptoms |
| XaCIs | All | Mild depression |
| XaCIt | All | Moderate depression |
| XaCIu | All | Severe depression |
| E0013 | All | Presenile dementia with depression |
| E0021 | All | Senile dementia with depression |

**Supplementary table S4.** Read codes used to identify, depression episodes.

| Read V2 | Term | |
|---|---|---|
| Code | ID | Description |
| E113. | All | Recurrent major depressive episode |
| E1130 | All | Recurrent major depressive episodes, unspecified |
| E1131 | All | Recurrent major depressive episodes, mild |
| E1132 | All | Recurrent major depressive episodes, moderate |
| E1133 | All | Recurrent major depressive episodes, severe, without mention of psychosis |
| E1134 | All | Recurrent major depressive episodes, severe, with psychosis |
| E1135 | All | Recurrent major depressive episodes, in partial or unspecified remission |
| E1136 | All | Recurrent major depressive episodes, in full remission |
| E1137 | All | Recurrent depression |
| E113z | All | Recurrent major depressive episode NOS |
| E2B1. | All | Chronic depression |
| Eu32A | All | [X]Recurrent major depressive episodes, severe, with psychosis, psychosis in remission |
| Eu33. | All | [X]Recurrent depressive disorder |
| Eu330 | All | [X]Recurrent depressive disorder, current episode mild |
| Eu331 | All | [X]Recurrent depressive disorder, current episode moderate |
| Eu332 | All | [X]Recurrent depressive disorder, current episode severe without psychotic symptoms |
| Eu333 | All | [X]Recurrent depressive disorder, current episode severe with psychotic symptoms |
| Eu334 | All | [X]Recurrent depressive disorder, currently in remission |
| Eu33y | All | [X]Other recurrent depressive disorders |
| Eu33z | All | [X]Recurrent depressive disorder, unspecified |
| Read CTV3 | Term | |
| Code | ID | Description |
| Xa0wV | All | Recurrent brief depressive disorder |
| XM1GC | All | Endogenous depression - recurrent |
| E1130 | All | Recurrent major depressive episodes, unspecified |
| E1131 | All | Recurrent major depressive episodes, mild |
| E1132 | All | Recurrent major depressive episodes, moderate |
| E1133 | All | Recurrent major depressive episodes, severe, without mention of psychosis |
| E1134 | All | Recurrent major depressive episodes, severe, with psychosis |
| XaX54 | All | Recurrent major depressive episodes, severe, with psychosis, psychosis in remission |
| E1135 | All | Recurrent major depressive episodes, in partial or unspecified remission |
| E1136 | All | Recurrent major depressive episodes, in full remission |
| E113z | All | Recurrent major depressive episode NOS |
| E1137 | All | Recurrent depression |
| E2B1. | All | Chronic depression |
| Eu331 | All | [X]Recurrent depressive disorder, current episode moderate |
| XE1Y1 | All | Recurrent major depressive episodes |

| | | [X]Recurrent depressive disorder, current episode severe without |
|---|---|---|
| XE1Zd | All | psychotic symptoms |
| | | [X]Recurrent depressive disorder, current episode severe with |
| XE1Ze | All | psychotic symptoms |
| XE1Zf | All | [X]Recurrent depressive disorder, unspecified |

**Supplementary table S5.** Read codes used to identify a diagnosis of recurrent major depression.

| Counselling | | |
|-------------|------|--------------------------------------------|
| Read V2 | Term | |
| Code | ID | Description |
| 67 | 11 | Counselling/health education |
| 671 | All | Counselling - general |
| 6712. | All | Counselling offered |
| 6714. | All | Counselling carried out |
| 6715. | All | Counselling by other agency |
| 6716. | All | Counselling of benefit |
| 6717. | All | Counselling of no benefit |
| 671Z. | All | Counselling - general NOS |
| 672 | All | Person counselled |
| 6721. | All | Patient counselled |
| 6722. | All | Family counselled |
| 673 | All | Person counselled by |
| 6731. | All | Counselled by a doctor |
| 6732. | All | Counselled by a nurse |
| 6733. | All | Counselled by a health visitor |
| 6735. | All | Counselled by a social worker |
| 6736. | All | Counselled by a counsellor |
| 6737. | All | Counselled by a vol. worker |
| 673Z. | All | Counselled by person NOS |
| 8M8 | All | Counselling requested |
| 9NJ1. | All | In-house counselling |
| 9NJR. | All | In-house counselling first appointment |
| 9NJT. | All | In-house counselling follow-up appointment |
| Read CTV3 | Term | in nouse counsening rollow up appointment |
| Code | ID | Description |
| X71Ec | All | Counselling |
| X71Ep | All | Coping strategy counselling |
| XaEC1 | All | Phobia counselling |
| XaD27 | All | Family counselling |
| 6779. | All | Psychological counselling |
| XaECG | All | Anxiety counselling |
| XaECF | All | Self-esteem counselling |
| XaI8j | All | Stress counselling |
| 672 | All | Person counselled |
| 6721. | All | Patient counselled |
| 6722. | All | Family counselled |
| XE1TI | All | Person counselled by |
| 6715. | All | Counselling by other agency |
| 6731. | All | Counselled by a doctor |
| 6732. | All | Counselled by a nurse |
| 6733. | All | Counselled by a health visitor |
| 6735. | All | Counselled by a social worker |

| 6736. | All | Counselled by a counsellor |
|---|---|---|
| 6737. | All | Counselled by voluntary worker |
| 673Z. | All | Counselled by person NOS |
| | All | <u> </u> |
| Xa07L | | Counselled by member of primary health care team |
| 9N2B. | All | Seen by counsellor |
| XaAS4 | All | Seen by mental health counsellor |
| XaBT1 | All | Refer to counsellor |
| XaAfJ | All | Referral to mental health counsellor |
| 9NJ1. | All | In-house counselling |
| XaLnp | All | In-house counselling first appointment |
| XaLnr | All | In-house counselling follow-up appointment |
| 671 | All | Counselling - general |
| 6712. | All | Counselling offered |
| 6714. | All | Counselling carried out |
| 6716. | All | Counselling of benefit |
| 6717. | All | Counselling of no benefit |
| 671Z. | All | Counselling - general NOS |
| XaA0d | All | Under care of counsellor |
| XaA0h | All | Under care of mental health counsellor |
| Cognitive Beh | | herapy |
| Read V2 | Term | Description |
| Code | ID | Description |
| 8G13. | All | Cognitive-behaviour therapy |
| 0.0420 | A 11 | [ C |
| 8G130 | All | Cognitive behavioural therapy parenting programme |
| 8G131 | All | CBTp - cognitive behavioural therapy for psychosis |
| 8G131<br>7L1a. | All<br>All | CBTp - cognitive behavioural therapy for psychosis Cognitive behavioural therapy |
| 8G131<br>7L1a.<br>7L1a0 | All<br>All<br>All | CBTp - cognitive behavioural therapy for psychosis Cognitive behavioural therapy Cognitive behavioural therapy by unidisciplinary team |
| 8G131<br>7L1a.<br>7L1a0<br>7L1a1 | All All All | CBTp - cognitive behavioural therapy for psychosis Cognitive behavioural therapy Cognitive behavioural therapy by unidisciplinary team Cognitive behavioural therapy by multidisciplinary team |
| 8G131<br>7L1a.<br>7L1a0<br>7L1a1<br>7L1ay | All All All All All | CBTp - cognitive behavioural therapy for psychosis Cognitive behavioural therapy Cognitive behavioural therapy by unidisciplinary team Cognitive behavioural therapy by multidisciplinary team Other specified cognitive behavioural therapy |
| 8G131 7L1a. 7L1a0 7L1a1 7L1ay 7L1az | All All All All All All All | CBTp - cognitive behavioural therapy for psychosis Cognitive behavioural therapy Cognitive behavioural therapy by unidisciplinary team Cognitive behavioural therapy by multidisciplinary team Other specified cognitive behavioural therapy Cognitive behavioural therapy NOS |
| 8G131 7L1a. 7L1a0 7L1a1 7L1ay 7L1az 8G510 | All | CBTp - cognitive behavioural therapy for psychosis Cognitive behavioural therapy Cognitive behavioural therapy by unidisciplinary team Cognitive behavioural therapy by multidisciplinary team Other specified cognitive behavioural therapy Cognitive behavioural therapy NOS Group cognitive behavioural therapy |
| 8G131 7L1a. 7L1a0 7L1a1 7L1ay 7L1az 8G510 8G15. | All | CBTp - cognitive behavioural therapy for psychosis Cognitive behavioural therapy Cognitive behavioural therapy by unidisciplinary team Cognitive behavioural therapy by multidisciplinary team Other specified cognitive behavioural therapy Cognitive behavioural therapy NOS Group cognitive behavioural therapy Computerised cognitive behavioural therapy |
| 8G131 7L1a. 7L1a0 7L1a1 7L1ay 7L1az 8G510 8G15. 8HIK. | All | CBTp - cognitive behavioural therapy for psychosis Cognitive behavioural therapy Cognitive behavioural therapy by unidisciplinary team Cognitive behavioural therapy by multidisciplinary team Other specified cognitive behavioural therapy Cognitive behavioural therapy NOS Group cognitive behavioural therapy |
| 8G131 7L1a. 7L1a0 7L1a1 7L1ay 7L1az 8G510 8G15. 8HIK. Read CTV3 | All Term | CBTp - cognitive behavioural therapy for psychosis Cognitive behavioural therapy Cognitive behavioural therapy by unidisciplinary team Cognitive behavioural therapy by multidisciplinary team Other specified cognitive behavioural therapy Cognitive behavioural therapy NOS Group cognitive behavioural therapy Computerised cognitive behavioural therapy Referral for cognitive behavioural therapy |
| 8G131 7L1a. 7L1a0 7L1a1 7L1ay 7L1az 8G510 8G15. 8HIK. Read CTV3 Code | All | CBTp - cognitive behavioural therapy for psychosis Cognitive behavioural therapy Cognitive behavioural therapy by unidisciplinary team Cognitive behavioural therapy by multidisciplinary team Other specified cognitive behavioural therapy Cognitive behavioural therapy NOS Group cognitive behavioural therapy Computerised cognitive behavioural therapy Referral for cognitive behavioural therapy Description |
| 8G131 7L1a. 7L1a0 7L1a1 7L1ay 7L1az 8G510 8G15. 8HIK. Read CTV3 Code Ub0qp | All | CBTp - cognitive behavioural therapy for psychosis Cognitive behavioural therapy Cognitive behavioural therapy by unidisciplinary team Cognitive behavioural therapy by multidisciplinary team Other specified cognitive behavioural therapy Cognitive behavioural therapy NOS Group cognitive behavioural therapy Computerised cognitive behavioural therapy Referral for cognitive behavioural therapy Description Cognitive and behavioural therapy |
| 8G131 7L1a. 7L1a0 7L1a1 7L1ay 7L1az 8G510 8G15. 8HIK. Read CTV3 Code Ub0qp XaABO | All | CBTp - cognitive behavioural therapy Cognitive behavioural therapy Cognitive behavioural therapy by unidisciplinary team Cognitive behavioural therapy by multidisciplinary team Other specified cognitive behavioural therapy Cognitive behavioural therapy NOS Group cognitive behavioural therapy Computerised cognitive behavioural therapy Referral for cognitive behavioural therapy Description Cognitive and behavioural therapy Cognitive - behaviour therapy |
| 8G131 7L1a. 7L1a0 7L1a1 7L1ay 7L1az 8G510 8G15. 8HIK. Read CTV3 Code Ub0qp XaABO Xad6J | All | CBTp - cognitive behavioural therapy for psychosis Cognitive behavioural therapy Cognitive behavioural therapy by unidisciplinary team Cognitive behavioural therapy by multidisciplinary team Other specified cognitive behavioural therapy Cognitive behavioural therapy NOS Group cognitive behavioural therapy Computerised cognitive behavioural therapy Referral for cognitive behavioural therapy Description Cognitive and behavioural therapy Cognitive - behaviour therapy Cognitive behavioural therapy |
| 8G131 7L1a. 7L1a0 7L1a1 7L1ay 7L1az 8G510 8G15. 8HIK. Read CTV3 Code Ub0qp XaABO Xad6J Xaaa6 | All | CBTp - cognitive behavioural therapy Cognitive behavioural therapy Cognitive behavioural therapy by unidisciplinary team Cognitive behavioural therapy by multidisciplinary team Other specified cognitive behavioural therapy Cognitive behavioural therapy NOS Group cognitive behavioural therapy Computerised cognitive behavioural therapy Referral for cognitive behavioural therapy Description Cognitive and behavioural therapy Cognitive - behaviour therapy Cognitive behavioural therapy Cognitive behavioural therapy Cognitive behavioural therapy Cognitive behavioural therapy for psychosis Cognitive behavioural therapy parenting programme |
| 8G131 7L1a. 7L1a0 7L1a1 7L1ay 7L1az 8G510 8G15. 8HIK. Read CTV3 Code Ub0qp XaABO Xad6J Xaaa6 XaQC0 | All | CBTp - cognitive behavioural therapy Cognitive behavioural therapy Cognitive behavioural therapy by unidisciplinary team Cognitive behavioural therapy by multidisciplinary team Other specified cognitive behavioural therapy Cognitive behavioural therapy NOS Group cognitive behavioural therapy Computerised cognitive behavioural therapy Referral for cognitive behavioural therapy Description Cognitive and behavioural therapy Cognitive - behaviour therapy Cognitive behavioural therapy Cognitive behavioural therapy for psychosis Cognitive behavioural therapy parenting programme Guided self help cognitive behavioural therapy |
| 8G131 7L1a. 7L1a0 7L1a1 7L1ay 7L1az 8G510 8G15. 8HIK. Read CTV3 Code Ub0qp XaABO Xad6J Xaaa6 XaQC0 XaKzQ | All | CBTp - cognitive behavioural therapy for psychosis Cognitive behavioural therapy Cognitive behavioural therapy by unidisciplinary team Cognitive behavioural therapy by multidisciplinary team Other specified cognitive behavioural therapy Cognitive behavioural therapy NOS Group cognitive behavioural therapy Computerised cognitive behavioural therapy Referral for cognitive behavioural therapy Description Cognitive and behavioural therapy Cognitive - behaviour therapy Cognitive behavioural therapy for psychosis Cognitive behavioural therapy parenting programme Guided self help cognitive behavioural therapy Computerised cognitive behavioural therapy |
| 8G131 7L1a. 7L1a0 7L1a1 7L1ay 7L1az 8G510 8G15. 8HIK. Read CTV3 Code Ub0qp XaABO Xad6J Xaaa6 XaQC0 XaKzQ Xa8I9 | All | CBTp - cognitive behavioural therapy Cognitive behavioural therapy by unidisciplinary team Cognitive behavioural therapy by multidisciplinary team Other specified cognitive behavioural therapy Cognitive behavioural therapy NOS Group cognitive behavioural therapy Computerised cognitive behavioural therapy Referral for cognitive behavioural therapy Pescription Cognitive and behavioural therapy Cognitive - behaviour therapy Cognitive behavioural therapy Cognitive behavioural therapy Cognitive behavioural therapy Cognitive behavioural therapy for psychosis Cognitive behavioural therapy parenting programme Guided self help cognitive behavioural therapy Computerised cognitive behavioural therapy Computerised cognitive behavioural therapy |
| 8G131 7L1a. 7L1a0 7L1a1 7L1ay 7L1az 8G510 8G15. 8HIK. Read CTV3 Code Ub0qp XaABO Xad6J Xaaa6 XaQC0 XaKzQ Xa8I9 XaM2I | All | CBTp - cognitive behavioural therapy Cognitive behavioural therapy by unidisciplinary team Cognitive behavioural therapy by multidisciplinary team Other specified cognitive behavioural therapy Cognitive behavioural therapy NOS Group cognitive behavioural therapy Computerised cognitive behavioural therapy Referral for cognitive behavioural therapy Description Cognitive and behavioural therapy Cognitive - behavioural therapy Cognitive behavioural therapy Cognitive behavioural therapy Cognitive behavioural therapy for psychosis Cognitive behavioural therapy parenting programme Guided self help cognitive behavioural therapy Computerised cognitive behavioural therapy Computerised cognitive behavioural therapy Cognitive behavioural therapy |
| 8G131 7L1a. 7L1a0 7L1a1 7L1ay 7L1az 8G510 8G15. 8HIK. Read CTV3 Code Ub0qp XaABO Xad6J Xaaa6 XaQC0 XaKzQ Xa8I9 | All | CBTp - cognitive behavioural therapy Cognitive behavioural therapy Cognitive behavioural therapy by unidisciplinary team Cognitive behavioural therapy by multidisciplinary team Other specified cognitive behavioural therapy Cognitive behavioural therapy NOS Group cognitive behavioural therapy Computerised cognitive behavioural therapy Referral for cognitive behavioural therapy Pescription Cognitive and behavioural therapy Cognitive - behaviour therapy Cognitive behavioural therapy Cognitive behavioural therapy for psychosis Cognitive behavioural therapy parenting programme Guided self help cognitive behavioural therapy Computerised cognitive behavioural therapy Computerised cognitive behavioural therapy |

| XaM2L | All | Cognitive behavioural therapy NOS |
|---|---|---|
| XaR2i | All | Referral to cognitive behavioural therapist |
| XaR5D | All | Referral for cognitive behavioural therapy |
| XaYgB | All | Referral for high intensity cognitive behavioural therapy |
| Psychotherap | | Referration high intensity cognitive behavioural dicrapy |
| Read V2 | Term | |
| Code | ID | Description |
| 8G | All | Psychotherapy |
| 8G1 | All | General psychotherapy |
| 8G10. | All | Psychotherapy - behavioural |
| 8G100 | All | Behavioural activation therapy |
| 8G101 | All | Dialectical behaviour therapy |
| 8G102 | All | Behavioural parent training |
| 8G11. | All | Psychotherapy - cognitive |
| 8G12. | All | Psychotherapy - psychodynamic |
| 8G120 | All | Short-term psychodynamic therapy |
| 8G121 | All | Dynamic interpersonal therapy |
| 8G122 | All | Focal psychodynamic therapy |
| 8G14. | All | Cognitive analytic therapy |
| 8G15. | All | Computerised cognitive behavioural therapy |
| 8G16. | All | Interpersonal psychotherapy |
| 8G18. | All | Cognitive stimulation therapy |
| 9NlK. | All | Seen by psychotherapist |
| 9NlK0 | All | Seen by trainee psychotherapist |
| 8ННТ. | All | Referral to psychotherapist |
| ZV57D | All | [V]Psychotherapy, not elsewhere classified |
| ZV673 | All | [V]Psychotherapy or other treatment for mental disorder follow-up |
| 8G9Z. | All | Other psychotherapy NOS |
| 8G9 | All | Other psychotherapy |
| Read CTV3 | Term | |
| Code | ID | Description |
| X71bp | All | Psychotherapy |
| XaaUO | All | Cognitive rehabilitation therapy |
| XaItc | All | Brief solution focused psychotherapy |
| Xa8IG | All | Psychoanalytic and psychodynamic therapy |
| Xa8IJ | All | Long-term exploratory psychotherapy |
| 3841. | All | Psychoanalysis |
| XaA8V | All | Generic psychoanalysis |
| XaA8W | All | Independent psychoanalysis |
| ХаА8Т | All | Kleinian psychoanalysis |
| XaA8U | All | Bion-based group psychoanalysis |
| XaA8X | All | Classical psychoanalysis |
| XaA8Y | All | Lacanian psychoanalysis |
| XaA8g | All | Group psychoanalysis |
| XaA8U | All | Bion-based group psychoanalysis |

| 384Z. | All | Psychological analysis NOS |
|-------|-----|---------------------------------------------------|
| Xa8IM | All | Jungian-based therapy |
| Xa8IN | All | Generic Jungian-based therapy |
| Xa8IP | All | Analytical psychology |
| Xa8IR | All | Long-term psychodynamic psychotherapy |
| XaA8Z | All | Developmental psychodynamic psychotherapy |
| XaA8c | All | Supportive expressive psychodynamic psychotherapy |
| XaA8d | All | Psychodynamic-interpersonal psychotherapy |
| XaEVq | All | Psychodynamic psychotherapy |
| Xad7C | All | Focal psychodynamic therapy |
| Xa8IR | All | Long-term psychodynamic psychotherapy |
| XaA8Z | All | Developmental psychodynamic psychotherapy |
| XaA8c | All | Supportive expressive psychodynamic psychotherapy |
| XaA8d | All | Psychodynamic-interpersonal psychotherapy |
| Xa8II | All | Short-term psychodynamic therapy |
| XaXuc | All | Dynamic interpersonal therapy |
| XaA9g | All | Specific task orientated psychotherapy |
| XE0iL | All | Psychotherapy/sociotherapy |
| 8G9Z. | All | Other psychotherapy NOS |
| 8G9 | All | Other psychotherapy |

**Supplementary table S6.** Read codes used to identify non-medication based treatments for depression or anxiety.

# Appendix 3

| <b>Medication class</b> | Medications |
|---|---|
| Medications for mental health conditions | |
| SSRIs and related medication | Venlafaxine, Bupropion, Duloxetine, Naltrexone,<br>Citalopram, Dapoxetine, Escitalopram, Fluoxetine,<br>Fluvoxamine, Paroxetine, Sertraline |
| TCAs | Amitriptyline, Clomipramine, Dosulepin, Doxepin,<br>Mianserin, Trazodone, Trimipramine, Imipramine,<br>Lofepramine, Nortriptyline |
| MAOIs | Tranylcypromine, Phenelzine, Isocarboxazid,<br>Moclobemide |
| Anxiolytic medications | Alprazolam, Chlordiazepoxide, Clobazam, Clonazepam,<br>Diazepam, Lorazepam, Oxazepam, Buspirone,<br>Meprobamate, Clomipramine, Clomethiazole |
| Medication for IBD | |
| Topical 5-ASA | Mesalazine, Sulfasalazine |
| Topical glucocorticoids | Budesonide, Hydrocortisone, Prednisolone |
| Oral 5-ASA | Balsalazide, Mesalazine, Olsalazine, Sulfasalazine |
| Oral glucocorticoids | Prednisolone, Cortisone, Dexamethasone,<br>Methylprednisolone, Beclomethasone, Betamethasone,<br>Budesonide, Deflazacort |
| Antimetabolites | Azathioprine, Mercaptopurine, Methotrexate |
| Biologic therapies | Adalimumab, Golimumab, Infliximab, Vedolizumab |

**Supplementary table S7.** Medications analysed by medication class. SSRI = selective serotonin reuptake inhibitors, TCA = tricyclic antidepressants, MAOI = monoamine oxidase inhibitors, 5ASA = 5-aminosalicylic acid.